CLINICAL TRIAL: NCT02248428
Title: Clarithromycin Plus CTd (Cyclophosphamide,Thalidomide and Dexamethasone)Regimen for Patients With Newly Diagnosed Multiple Myeloma:a Phase 3 , Multicenter,Randomized, Open-Label Trial.
Brief Title: Clarithromycin Plus CTd Regimen for Patients With Newly Diagnosed Multiple Myeloma
Acronym: CTd
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Yongping Zhai, Department of hemotology, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAB20140324
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; Clarithromycin; CTd
MeSH Terms: conditions — Multiple Myeloma | interventions — Clarithromycin; Thalidomide; Cyclophosphamide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BiCTd regimen (Experimental): Induction and consolidation therapy: BiCTd regimen for 8 cycles. Patients received Clarithromycin 500 mg orally on days 1-28,thalidomide 100-200mg orally on days d1-28, dexamethasone 40mg orally on days on 1,8,15,22, and cyclophosphamide 300mg/m^2 intravenously on day 1-3. Cycles were repeated every 28 days.
  Maintenance therapy:CP regimen (cyclophosphamide 200 mg orally on days 1-14 and prednisone 30mg twice daily orally on days 1-7,repeated every 28 days) until disease progression.
  If efficacy <PR after 4 cycles of induction or disease progression at anytime，patients will be quitted.
  Interventions: Drug: Clarithromycin; Drug: Thalidomide; Drug: Cyclophosphamide; Drug: Dexamethasone
- CTd regimen (Active Comparator): Induction and consolidation therapy: CTd regimen for 8 cycles. Patients received thalidomide 100-200mg orally on days d1-28, dexamethasone 40 mg orally on days on 1,8,15,22, and cyclophosphamide 300 mg/m^2 intravenously on day 1-3. Cycles were repeated every 28 days.
  Maintenance therapy:CP regimen (cyclophosphamide 200 mg orally on days 1-14 and prednisone 30mg twice daily orally on days 1-7,28 Days per Cycle) until disease progression.
  If efficacy <PR after 4 cycles of induction or disease progression at anytime，patients will be quitted.
  If no further reduction in the serum and urine M protein in the next cycle，patients may cross over to BiCTd regimen.
  Interventions: Drug: Thalidomide; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Clarithromycin — 500mg orally daily on days 1-28,repeated every 28 days
  Other Names: Abbott- 56268; Biaxin; CLARITH
  Arms: BiCTd regimen
Drug: Thalidomide — Thalidomide 100-200mg orally per night on days 1-28,repeated every 28 days
  Other Names: Distaval; Thalomid
Drug: Cyclophosphamide — 300mg/m^2 intravenously daily on day 1-3,repeated every 28 days
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune
Drug: Dexamethasone — 40 mg orally weekly on days 1,8,15,22,repeated every 28 days
  Other Names: Decadron; Aeroseb-Dex; Decaderm; DM; DXM

SUMMARY:
Due to economic reasons, thalidomide is still widely used as a first line drug for Multiple Myeloma patients in China. However,the efficacy of CTd is still lower than the therapeutic regimens with new drugs. Clarithromycin may have partly efficacy in association with steroids and thalidomide for Multiple Myeloma patients. This multicenter, randomized, phase 3 clinical trial is proposed to explore whether clarithromycin could potentiate responsiveness of CTd (Cyclophosphamide, Thalidomide and Dexamethasone) regimen in Newly Diagnosed Multiple Myeloma patients. The trial will also evaluate the side effects caused by the combination of these drugs.

DETAILED DESCRIPTION:
This phase III,randomized controlled trial will enroll 130(65 each arm) newly diagnosed patients with active disease from 4 medical centers in East China.

The participants are randomly equally selected to receive BiCTd regimen arm or CTd regimen arm. The treatment consists of eight induction and consolidation therapy followed by maintenance therapy.

BiCTd(Clarithromycin, Cyclophosphamide, Thalidomide and Dexamethasone) regimen arm：

Induction and consolidation Phase:

All patients will also receive aspirin 100mg PO QD while receiving BiCTd. Aspirin will continue through maintenance.

Clarithromycin 500 mg orally daily on days 1-28,thalidomide 100-200mg orally on days d1-28, dexamethasone 40 mg orally on days on 1,8,15,22, and cyclophosphamide 300 mg/m^2 intravenously on day 1-3. Eight Cycles were repeated every 28 days.

If efficacy <PR after 4 cycles of induction， or disease progression at anytime，patients will be quitted.

Maintenance Therapy:

Patients who complete the induction and consolidation regimen could be started on maintenance therapy as follows: Maintenance with CP (cyclophosphamide 200 mg orally on days 1-14 and prednisone 30mg twice daily orally on days 1-7,repeated every 28 days) regimen until disease progression.

CTd regimen arm：

Induction and consolidation Phase:

All patients will also receive aspirin 100mg PO QD while receiving CTd. Aspirin will continue through maintenance.

Thalidomide 100-200mg orally on days d1-28, dexamethasone 40 mg orally on days on 1,8,15,22, and cyclophosphamide 300 mg/m^2 intravenously on day 1-3. Eight Cycles were repeated every 28 days.

If efficacy <PR after 4 cycles of induction， or disease progression at anytime，patients will be quitted.

If no further reduction in the serum and urine M protein in the next cycle，patients may cross over to BiCTd regimen.

Maintenance Therapy:

Patients who complete the induction and consolidation regimen could be started on maintenance therapy as follows: Maintenance with CP (cyclophosphamide 200 mg orally on days 1-14 and prednisone 30mg twice daily orally on days 1-7,repeated every 28 days) regimen until disease progression Then, patients will be followed up for 24 months after chemotherapy. The investigators will record all the laboratory and clinical investigations to assess response at different points of the study. We also assess adverse events (AEs), as graded according to NCI-Common Toxicity Criteria for Adverse Effects (CTCAE) Version 4.0.Response categories were based on the International Myeloma Working Group uniform response criteria.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Diagnosed with active multiple myeloma
* Previously untreated
* Karnofsky performance status(KPS) ≥50（KPS<50 will be allowed if related to bony disease）
* New York Heart Association(NYHA) functional ≤class III

Exclusion Criteria:

* Hypersensitivity to clarithromycin or any of its excipients, erythromycin, or any of the macrolide antibiotics;
* Concomitant administration of cisapride, pimozide, astemizole, terfenadine, ergotamine or dihydroergotamine, simvastatin, lovastatin, and atorvastatin;
* A history of cholestatic jaundice/hepatic dysfunction associated with prior use of clarithromycin.
* Impaired renal function,Creatinine ≥221umol/L；
* Pregnant or breast feeding females.
* Any condition which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-04; Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Very Good Partial Remission (VGPR) or Better | up to 4 months
  Quality of response: % Complete Response (CR) + Very Good Partial Remission (VGPR) to induction BiCTd or CTd as assessed using International Myeloma Working Group Response Definitions. Very Good Partial Remission (VGPR): Detectable serum and urine M component on immunofixation but not on electrophoresis or 90% or greater reduction in serum M protein with less than 100 mg/24 h of urinary M protein. Complete Remission (CR): The presence of less than 5% bone marrow plasmacytosis and the disappearance of all evidence of serum and urine M-components on electrophoresis as well as by immunofixation. In addition, soft tissue plasmacytoma must have disappeared.

SECONDARY OUTCOMES:
Median Progression Free Survival (PFS) in months | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 Months
  PFS: Time from study entry to progression/relapse or death from study entry to death of any cause, assessed using International Myeloma Working Group Response Definitions. Progressive Disease (PD): One of the following criteria must be met: a. Increase of 25% or greater in serum M protein (absolute increase greater or equal to 0.5g/dl); b. Increase of 25% or greater in urine M protein (absolute increase greater than 200 mg/24h); c. Increase of 25% or greater in the difference between the involved and uninvolved free light chain (absolute increase greater than 10 mg/dl); d. Increase of 25% or greater in bone marrow plasma cell percentage (absolute percent greater than 5% in case the patient was in CR and 10% otherwise); i.e. Definite development of new bone lesions or soft tissue plasmacytomas, or increase in the size of existing plasmacytomas by greater or equal to 25%. Development of hypercalcemia (serum calcium > 11.5 mg/dl) attributable only to the plasma cell dyscrasia.
2 Year Overall Survival (OS) Rate | up to 24 months
  Percentage of participants with Overall Survival in response to BiCTd or CTd in newly diagnosed multiple myeloma patients with active disease. Overall survival is time from study entry to death of any cause.
Number of participants with adverse events | up to 48 months
  Adverse events (AEs) were graded according to NCI-CTCAE Version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Yongping Zhai, doctor, Study Chair — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China